CLINICAL TRIAL: NCT02982486
Title: A Phase II Single Arm Study Assessing Efficacy & Safety of Nivolumab Plus Ipilimumab in Nonresectable/Metastatic Sarcoma and Endometrial Carcinoma Patients With Somatic Deficient MMR as a Selection Tool
Brief Title: A Phase II of Nivolumab Plus Ipilimumab in Non-resectable Sarcoma and Endometrial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Daniela Katz M.D, M.D, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0239/16
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Soft Tissue Sarcoma; Bone Sarcoma; Chondrosarcoma; Gastrointestinal Stromal Sarcoma; Ewing's Tumor Metastatic; Ewing's Tumor Recurrent; Osteosarcoma; Desmoplastic Small Round Cell Tumor
Keywords: nivolumab; ipilimumab; immunotherapy; PD-1 inhibitor; sarcoma
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Chondrosarcoma; Gastrointestinal Stromal Tumors; Osteosarcoma; Desmoplastic Small Round Cell Tumor | interventions — Ipilimumab; Nivolumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab and ipilimumab (Experimental): Nivolumab 240 mg IV every 2 weeks plus Ipilimumab 1 mg/m2 IV every 6 weeks
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 1 mg/kg every 6 weeks
  Other Names: anti CTLA4
Drug: Nivolumab — Ninolumab 240 mg IV every 2 weeks
  Other Names: Anti PD-1

SUMMARY:
The purpose of this study is to determine whether nivolumab plus ipilimumab are effective and safe in the treatment of sarcoma and endometrial carcinoma patients with somatic deficient MMR as a selection tool.

DETAILED DESCRIPTION:
The expected duration of this study is 36 months (18 months accrual period and 18 month follow up period). Enrollment into the screening or treatment phase of the study will be stopped when the actual subject numbers have been achieved.

This single arm single institution, open label, prospective, phase II trial will evaluate the efficacy and safety of Nivolumab 240 mg IV every 2 weeks plus ipilimumab 1 mg/kg every 6 weeks in patients with nonresectable/metastatic sarcoma or endometrial carcinoma with somatic deficient MMR as a selection tool.patients. Number of patients in the study will reflect the reconciliation between statistical requirements and incidence.

Treatment will continue until disease progression, development of unacceptable toxicity, noncompliance or withdrawal of consent by the patient or investigator decision.

All screening requirements must be completed within 28 days of the visit (except for Patients will be examined on cycle 1 day-1 and every 2 weeks, including complete blood count (CBC) and chemistry, until disease progression. CT/MRI imaging (contrast) will be performed every 6 weeks for response evaluation for the first 48 weeks and every 12 weeks thereafter. Clinical benefit as well as individual categories of response (complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) will be determined using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST). Response duration endpoints, including median PFS, PFS at 12 and 24 weeks and OS will be assessed using the Kaplan-Meier method. Toxicity (AEs) will be recorded using the NCI- Common Toxicity Criteria for Adverse Effects v 4.03 (NCI-CTCAE). Screening procedures will include immunostaining for MLH1, MSH2, MSH6 and PMS2 all performed on formalin fixed paraffin embedded (FFPE) tissue sections. In addition tumor DNA, extracted from FFPE tissue (after choosing optimal area by a Pathologist), will be submitted to FoundationOne for a later exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will sign the informed consent form before the initiation of any study procedure.
2. Males and Females, 18 years or older
3. Patients must have a FFPE tumor block, one representative hematoxylin and eosin (H&E) and 20 unstained sarcoma/endometrial carcinoma tissue slides available for submission to pathology review; this step is mandatory prior to registration to confirm eligibility.
4. Tumors must immune-stain negatively to one or more of the following proteins: MLH1, MSH2, MSH6 and PMS2
5. Patients must have histologically confirmed bone or soft tissue sarcoma by pathology review or a diagnosis of FIGO grade 3 endometrioid cancer, serous, clear cell, or mixed high grade endometrial cancer.
6. Measurable disease of sarcoma or endometrial carcinoma defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan or MRI, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam by RECIST 1.1.
7. Locally advanced non-operable or metastatic disease
8. >= 1 prior systemic therapy for sarcoma or endometrial carcinoma, including adjuvant systemic therapy
9. No treatment with biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy =< 21 days before study registration
10. Eastern Cooperative Oncology Group ECOG performance status 0 or 1
11. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to first drug dose

    * WBC ≥ 2000/μL
    * Neutrophils ≥ 1500/μL
    * Platelets ≥ 100 x103/μL
    * Hemoglobin > 9.0 g/dL
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

      * Female CrCl = (140 - age in years) x weight in kg x 0.85

        72 x serum creatinine in mg/dL
      * Male CrCl = (140 - age in years) x weight in kg x 1.00

        72 x serum creatinine in mg/dL
    * AST/ALT ≤ 3 x ULN
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
    * Serum electrolytes: baseline serum potassium > 3.5 mmol/L (potassium supplementation may be given to restore the serum potassium above this level prior to study entry)
    * Thyroid stimulating hormone (TSH) within normal limits (WNL); supplementation is acceptable to achieve a TSH WNL; in patients with abnormal TSH if free T4 is normal and patient is clinically euthyroid, patient is eligible
12. Patients should have resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE, version 4.0, grade 1 or less
13. Patients may be re-screened and re-enrolled in the study if they failed screening or were enrolled but did not receive study drugs in this case they will have to sign a new informed concent form.
14. Palliative (limited-field) radiation therapy is permitted, if all of the following criteria are met:

    * Repeat imaging demonstrates no new sites of bone metastases.
    * The lesion being considered for palliative radiation is not a target lesion.
15. A negative pregnancy test (a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG)) done =< 7 days prior to the start of study drug.
16. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
17. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab
18. Women must not be breastfeeding
19. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception

Exclusion Criteria:

1. Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
2. Have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
3. FIGO grade 1 or 2 endometrioid cancer.
4. Have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
5. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of nivolumab/ipilimumab or has not recovered (i.e., to ≤ grade 1 or baseline) from adverse events due to a previously administered agent. Note, subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note, if a subject received major surgery, she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. No known or suspected allergy to nivolumab or study drug components and no history of severe hypersensitivity reaction to any monoclonal antibody
7. Active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
8. As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
9. Have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
10. Have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
11. Known active pulmonary disease with hypoxia defined as:

    Oxygen saturation < 85% on room air or Oxygen saturation < 88% despite supplemental oxygen
12. Pregnant and nursing women
13. Eastern Cooperative Oncology Group (ECOG) performance status 3-4
14. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Response to therapy as evaluated by RECIST 1.1 | 36 months
  complete and partial response

SECONDARY OUTCOMES:
Median Progression-free survival (PFS) | 36 months
  PFS will be computed from the date of start of treatment to the first documented date of progression or the date of death, due to any cause assessed by investigator.
Progression-free survival (PFS) assessed at 12 weeks | 12 weeks
  PFS will be computed from the date of start of treatment to week 12 as assessed by investigator.
Progression-free survival (PFS) assessed at 24 weeks | 24 weeks
  PFS will be computed from the date of start of treatment to week 24 as assessed by investigator
overall survival | 36 months
  will be computed from the date of start of treatment to the date of death, due to any cause. Patients alive or lost for follow-up at the time of the analysis will be censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Katz, M.D, Principal Investigator — Assaf-Harofeh Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255